CLINICAL TRIAL: NCT06202014
Title: Phase II Study of Concurrent Radiotherapy With Envafolimab and Capecitabine in Locally Advanced Pancreatic Cancer
Brief Title: Phase II Study of Concurrent Radiotherapy With Envafolimab and Capecitabine in LAPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, BO CHEN, Associate Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4325
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer; Radiotherapy; Envafolimab; Capecitabine
Keywords: pancreatic cancer; envafolimab; capecitabine; radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — envafolimab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concurrent Radiotherapy With Envafolimab and Capecitabine (Experimental): Concurrent radiotherapy with envafolimab and capecitabine, post-adjuvant envafolimab and capecitabine for locally advanced pancreatic cancer
  Interventions: Radiation: concurrent radiotherapy with envafolimab and capecitabine

INTERVENTIONS:
Radiation: concurrent radiotherapy with envafolimab and capecitabine — Eligibility patients will receive intensity-modulated radiotherapy(IMRT)or volumetric modulated arc therapy(VMAT) to pancreatic lesions,metastatic lymph nodes and high-risk lymphatic drainage areas,concurrent with and followed by envafolimab and capecitabine.Concurrent and sequential dose of envafolimab is 200mg subcutaneous injection weekly.Capecitabine is with a concurrent and sequential dose of 500-800 mg/m2 bid po , taken orally for 2 weeks and stopped for 1 week (standard concurrent dose is 800 mg/m2 bid po , but for patients ≥70 years of age, 500 mg/m2 bid po depending on physical status ) until progression or intolerance.

SUMMARY:
This is a single-arm prospective phase II clinical trial to investigate the efficacy and safety of concurrent radiotherapy with envafolimab and capecitabine in locally advanced pancreatic cancer.Eligibility patients will receive intensity-modulated radiotherapy(IMRT)or volumetric modulated arc therapy(VMAT) to pancreatic lesions,metastatic lymph nodes and high-risk lymphatic drainage areas,concurrent with and followed by envafolimab and capecitabine.

DETAILED DESCRIPTION:
This is a single-arm prospective phase II clinical trial to investigate the efficacy and safety of concurrent radiotherapy with envafolimab and capecitabine in locally advanced pancreatic cancer.Primary enrollment criteria is locally advanced non-resectable pancreatic cancer without systemic metastases other than retroperitoneal lymph nodes.Eligibility patients will receive intensity-modulated radiotherapy(IMRT)or volumetric modulated arc therapy(VMAT) to pancreatic lesions,metastatic lymph nodes and high-risk lymphatic drainage areas,concurrent with and followed by envafolimab and capecitabine.Concurrent and sequential dose of envafolimab is 200mg subcutaneous injection weekly.Capecitabine is with a concurrent and sequential dose of 500-800 mg/m2 bid po , taken orally for 2 weeks and stopped for 1 week (standard concurrent dose is 800 mg/m2 bid po , but for patients ≥70 years of age, 500 mg/m2 bid po depending on physical status ) until progression or intolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-90 years old.
2. Pancreatic cancer diagnosed by histology or cytology.
3. Locally or regionally advanced non-resectable pancreatic cancer without systemic metastases other than retroperitoneal lymph nodes.
4. Patients who have not received prior systemic chemotherapy or who have progressed on first-line therapy.
5. At least one measurable lesion (≥10 mm long diameter on CT scan for tumor lesions and ≥15 mm short diameter on CT scan for lymph node lesions according to RECIST 1.1 criteria).
6. ECOG score: 0-1.
7. Expected survival ≥ 3 months.
8. Normal function of major organs, meeting the following criteria:
9. Criteria for routine blood tests need to be met (no blood and blood products transfusion within 14 days):

   1. ANC ≥ 1.5×10^9/L
   2. PLT ≥80×10^9/L
10. Biochemical tests need to meet the following criteria:

    1. TBIL<1.5 ULN
    2. ALT and AST < 2.5ULN and in patients with liver metastases < 5ULN
    3. Serum Cr ≤ 1.25ULN or endogenous creatinine clearance > 45 ml/min (Cockcroft-Gault formula) 11).Subjects voluntarily enrolled in this study and signed an informed consent form, were compliant and cooperated with the follow-up.

Exclusion Criteria:

1. Presence of any active autoimmune disease or history of autoimmune disease in the subject.
2. Allergy to study-used medications.
3. Subjects who are on immunosuppressive, or systemic, or absorbable topical hormone therapy for immunosuppression (dose >10mg/day prednisone or other equipotent hormone) and who continue to be on it within 2 weeks prior to enrollment.
4. Class III-IV cardiac insufficiency according to NYHA criteria, or cardiac ultrasound suggesting left ventricular ejection fraction (LVEF) <50%.
5. Those with abnormal coagulation function (INR>1.5,APTT>1.5 ULN) and bleeding tendency.
6. prolonged unhealed wounds or fractures; major surgical procedures or severe traumatic injuries, fractures or ulcers within 4 weeks.
7. Subjects with congenital or acquired immune deficiency (e.g., HIV-infected individuals), or active hepatitis (Hepatitis B reference: HBV DNA test value exceeding the upper limit of normal, Hepatitis C reference: HCV viral titer or RNA test value exceeding the upper limit of normal).
8. Subject has received other prior PD-1 antibody immunotherapy or other immunotherapy targeting PD-1 or PD-L1.
9. Known existing hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophiliacs, coagulation disorders, thrombocytopenia, hypersplenism, etc.) or events of arterial or venous thrombosis in the last 6 months (up to the first medication use of envafolimab ).
10. Subjects with active infection or unexplained fever >38.5 degrees Celsius during screening and prior to the first dose.
11. Patients with central nervous system metastases;
12. Subjects who have had a live bacterial vaccine or live attenuated vaccine vaccine within 30 days prior to the first dose of study treatment.
13. Subjects with previous or concurrent other malignant tumors.
14. Women who are pregnant or breastfeeding.
15. Those with a history of psychotropic substance abuse that cannot be abstained from or patients with psychiatric disorders.
16. Patients with concomitant illnesses that, in the judgment of the investigator, seriously jeopardize patient safety or interfere with the patient's ability to complete the study.
17. Those who are not suitable for inclusion in the judgment of the investigator.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 1-3 months after radiotherapy
  Overall Response Rate (ORR) was defined as the total of CR (Complete Response) and PR (Partial Response). CR and PR were assessed by independent reviewers according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR evaluated in 1 to 3 months after the completion of radiotherapy.

SECONDARY OUTCOMES:
PFS | up to 24 months
  Progress free survival
OS | up to 24 months
  Overall Survival (OS) was defined as the duration from the date of patient recruited to the date of death with any reason
DCR | up to 24 months
  Complete response(CR)and partial response(PR)
DoR | up to 24 months
  During of response
Incidence of grade 3 and above adverse events | up to 24 months
  Adverse events was evaluated during received protocol therapy according to the NCI Common Terminology Criteria for Adverse Events 4.03(CTCAE 4.03).

CONTACTS AND LOCATIONS:
Locations (1):
- Bo Chen, Beijing, Beijing Municipality, China